CLINICAL TRIAL: NCT03269721
Title: Determinants of Altered Brain Structure and Function in Smokers With COPD-Related Lung Pathophysiology
Brief Title: COPD-Related Physiology and the Brain
Status: Completed | Type: Observational
Sponsor: Karin Hoth (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor-Investigator, Karin Hoth, Professor, University of Iowa
Organization: University of Iowa (Other)
Other Study IDs: 201404738; 1R01HL134822-01 (NIH)
Record Dates: First submitted 2017-08-30; First posted 2017-09-01 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Pulmonary Disease, Chronic Obstructive (COPD); Cognitive Impairment
Keywords: Cognition; Pulmonary; COPD; Lung
MeSH Terms: conditions — Lung Diseases; Pulmonary Disease, Chronic Obstructive; Cognitive Dysfunction | interventions — Neuropsychological Tests; Blood Gas Analysis; Carbon Monoxide; Walk Test

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stored blood samples may be used to evaluate additional biomarkers. These future studies may provide additional information that will be helpful in understanding COPD and its comorbidities. If consent is given, samples may also be used for potential genetic research.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Never Smoker: Neuropsychological Assessment, Spirometry, Arterial Blood Gas, Diffusion Capacity of the Lung for Carbon Monoxide, 6 Minute Walk test, Systemic Vascular Measures, Blood Biomarkers, Symptom Questionnaire Measures, Brain MRI
  Interventions: Behavioral: Neuropsychological Assessment; Procedure: Spirometry; Procedure: Arterial Blood Gas; Procedure: Diffusion Capacity of the Lung for Carbon Monoxide; Diagnostic Test: 6 Minute Walk Test; Procedure: Systemic Vascular Measures; Biological: Blood Biomarkers; Behavioral: Symptom Questionnaire Measures; Procedure: Brain MRI
- Smoker/Past smoker-No Airflow Limitation: Neuropsychological Assessment, Spirometry, Arterial Blood Gas, Diffusion Capacity of the Lung for Carbon Monoxide, 6 Minute Walk test, Systemic Vascular Measures, Blood Biomarkers, Symptom Questionnaire Measures, Brain MRI
  Interventions: Behavioral: Neuropsychological Assessment; Procedure: Spirometry; Procedure: Arterial Blood Gas; Procedure: Diffusion Capacity of the Lung for Carbon Monoxide; Diagnostic Test: 6 Minute Walk Test; Procedure: Systemic Vascular Measures; Biological: Blood Biomarkers; Behavioral: Symptom Questionnaire Measures; Procedure: Brain MRI
- Smoker/Past smoker-W/Airflow Limitation: Neuropsychological Assessment, Spirometry, Arterial Blood Gas, Diffusion Capacity of the Lung for Carbon Monoxide, 6 Minute Walk test, Systemic Vascular Measures, Blood Biomarkers, Symptom Questionnaire Measures, Brain MRI
  Interventions: Behavioral: Neuropsychological Assessment; Procedure: Spirometry; Procedure: Arterial Blood Gas; Procedure: Diffusion Capacity of the Lung for Carbon Monoxide; Diagnostic Test: 6 Minute Walk Test; Procedure: Systemic Vascular Measures; Biological: Blood Biomarkers; Behavioral: Symptom Questionnaire Measures; Procedure: Brain MRI

INTERVENTIONS:
Behavioral: Neuropsychological Assessment — Assessments include: Paper and pencil computerized measures of Memory, Language, Visuospatial Function, Executive Functioning-Processing Speed, and Attention
Procedure: Spirometry — Pre and post bronchodilator spirometry will be administered according to the American Thoracic Society (ATS) guidelines.
Procedure: Arterial Blood Gas — Radial artery blood sample will be collected to measure gas exchange hemoglobin; arterial oxygen and carbon dioxide will be examined as potential covariates.
Procedure: Diffusion Capacity of the Lung for Carbon Monoxide — For measurement of gas exchange in the lung. DLCO adjusted for hemoglobin will be the primary variable of interest and will be examined as a potential covariate.
  Other Names: (DLCO)
Diagnostic Test: 6 Minute Walk Test — Distance walked in 6 minutes will be the primary outcome.
  Other Names: 6MWT
Procedure: Systemic Vascular Measures — Carotid artery ultrasound, pulse wave velocity, brachial artery endothelium-dependent flow mediated dilation and endothelium-independent dilation will be measured.
Biological: Blood Biomarkers — High sensitivity C-reactive protein (hs-CRP), and fibrinogen will be used as indicators of systemic inflammation, complete blood count with differential (CBC with diff) will be obtained to rule out acute infection as a cause of inflammation.
Behavioral: Symptom Questionnaire Measures — M.I.N.I Screen 7.0.0, Beck Depression Inventory-II (DBI-II), State Trait Anxiety Inventory (STAI), COPD Assessment Test (CAT), St. George's Respiratory Questionnaire (SGRQ), MMRC Dyspnea Scale (MMRC), Berlin Questionnaire
Procedure: Brain MRI — Primary neuroimaging outcomes of interest are white matter structural integrity

SUMMARY:
COPD is the third leading cause of combined morbidity, disability, and mortality in the United States and is often associated with cognitive impairment. The goal of the proposed project is to examine novel pulmonary and vascular physiological mechanisms that contribute to structural brain abnormalities and cognitive dysfunction early in the course of COPD. The project will generate information to ultimately inform the development of interventions to delay or prevent cognitive dysfunction.

DETAILED DESCRIPTION:
Chronic Obstructive Pulmonary Disease (COPD) is the 3rd leading cause of morbidity and mortality in the US with increasing prevalence in older adults. The impact of COPD on the brain is an area of expanding research interest. A staggering 40-60% of patients with COPD have cognitive impairments including deficits in executive functioning (e.g., decision making), processing speed, and memory. Intact cognition is critical for independently managing daily tasks (e.g., medication and money management). Since there are currently no treatments to fully reverse cognitive impairment once it is present, preventing and delaying onset is essential. Given the high prevalence of COPD, understanding how COPD confers an increased risk for cognitive impairment should be a top public health priority. There is an urgent need to identify potentially modifiable physiological characteristics of individuals with early COPD-related pathophysiology who are at risk of developing brain abnormalities. The earliest changes that occur in COPD are driven by an enhanced chronic inflammatory response that includes small airway disease in the lung and vascular abnormalities. COPD-related lung pathophysiology can be measured continuously and is separable from amount of smoking. These physiological changes are often present in individuals who do not meet traditional criteria for COPD diagnosis and have not yet manifested significant clinical symptoms. We propose that chronic smokers who are susceptible to COPD and show evidence of COPD-related lung pathophysiology on lung CT also experience vascular dysfunction (particularly central artery stiffness) that contributes to structural brain abnormalities and cognitive impairment. The proposed project will: 1) model the effects of novel physiological mechanisms on the brain in COPD, 2) focus on changes in brain structure and function early in the development of COPD by including smokers who have evidence of early COPD-related lung pathophysiology but do not meet traditional criteria for COPD, and 3) utilize advanced technology to assess the lung (lung CT) and brain (MRI). We will recruit participants with existing lung CT from ongoing NIH projects to complete pulmonary and vascular measures, cognitive assessment, and brain MRI. The project is highly multidisciplinary and leverages unique resources at the University of Iowa including the Institute for Clinical and Translational Science, the Translational Human Vascular Physiology Lab, the Iowa Neuroimaging Consortium, and the Iowa Comprehensive Lung Imaging Center.

ELIGIBILITY:
Inclusion Criteria:

Age 30-85, > 8th grade education, Normal/corrected hearing and vision, English Speaker, Ability to comfortably lie flat for 1 hour.

Exclusion Criteria:

Other concomitant respiratory disorder other than asthma (e.g., cystic fibrosis), Use of antibiotics or steroids for a COPD exacerbation within the past month, Use of 24-hour oxygen, Pregnancy or suspected pregnancy, Uncontrolled cancer within the last 5 years, Radiation therapy to the chest, Lung surgery (LVRS, transplant, lobectomy), Lung cancer known or suspected, Eye surgery in the last 3 months, Pulmonary Hypertension, Insulin-dependent diabetes, Inability to use albuterol, Chest or abdominal surgery in the past 3 months, Heart attack in the last 3 months, Hospitalization for any heart problem in the past month, Prior neurological condition (e.g., stroke, epilepsy, head injury with >15 mins. loss of consciousness), Previous diagnosis of dementia or learning disability, Major comorbid medical conditions with known cognitive effects (e.g., renal failure, HF), Psychotic disorder, bipolar disorder, current substance use disorder other than tobacco use, Change in psychiatric medication in last month, Claustrophobia, Metal object in body that may interfere with neuroimaging.

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from the Iowa COPD research registry, which includes participants from several NIH funded studies with quantitative lung imaging obtained in the Iowa Comprehensive Lung Imaging Center.
Sampling Method: Non-Probability Sample
Enrollment: 170 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
White matter (WM) structural integrity from brain magnetic resonance imaging (MRI) | At the end of data collection in 2024
  Fractional anisotropy from diffusion weighted imaging will be the primary WM measure
Neuropsychological test performance: average executive functioning-processing speed domain summary score | At the end of data collection in 2024
  The domain summary score represents the average of the norm referenced standardized scores for the following measures: Trail Making Test Part B, Controlled Oral Word Association, Stroop Color Word Test Interference Score, and WAIS-IV (Wechsler Adult Intelligence Scale IV) Coding

CONTACTS AND LOCATIONS:
Overall Officials: Karin F Hoth, PhD, Principal Investigator — University of Iowa Department of Psychiatry
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No